

# STATISTICAL REPORTING AND ANALYSIS PLAN

# CLINICAL STUDY TO MEASURE THE IMPACT OF FORTIFIED MALT BASED FOOD ON IMMUNITY OUTCOMES IN SCHOOL CHILDREN

**Protocol Number: 204477** 

Phase: N/A

Property of GSK Consumer Healthcare
Confidential
May not be used, divulged, published or otherwise disclosed
without the consent of GSK

Template Version Effective: 15-Jul-2017


# **Document History**

| Document | Version Date | Summary of Changes (New analysis or Change in planned analysis) |
|---|---|---|
| Original Analysis Plan | 27-June -2018 | Not applicable (N/A) |
| Amendment 1 | 2-November-2018 | <ol> <li>For all ANCOVA analyses, "cluster (school)" will be included as a random effect instead of a fixed effect. Handling "cluster" as random effect would avoid over-parametrisation and would allow for intracluster correlation.</li> <li>Present the estimate of the intra cluster correlation in the ANCOVA tables. Adjusting for the intracluster correlation is necessary for a valid analysis.</li> <li>Implementation of comments received during dry-run process.</li> <li>Creation of additional corresponding descriptive statistics tables for exploratory ANCOVA tables.</li> <li>Removal of raw outputs in section 16.1.9 with no corresponding ANCOVA tables in section 14.2.</li> <li>Replacing originally planned figures with corresponding tables.</li> </ol> |

# **Table of contents**

| | Docui | ment Histo | ory | 2 |
|---|---|---|---|---|
| | Table | of conten | ts | 3 |
| | Abbreviations5 | | | |
| 1 | Sumn | nary of Ke | ey Protocol Information | 7 |
| | 1.1 | Study D | esign | 7 |
| | 1.2 | Study O | bjectives | 9 |
| | 1.3 | Treatme | nts | 11 |
| | 1.4 | Sample | Size Calculation | 11 |
| 2 | Plann | ed Analys | es | 12 |
| | 2.1 | Interim | Analysis | 12 |
| | 2.2 | Final Ar | nalyses | 12 |
| 3 | Consi | derations | for data analyses and Data Handling Conventions | 13 |
| | 3.1 | Baseline | Definition | 13 |
| | 3.2 | Subgrou | ps/Stratifications | 13 |
| | 3.3 | Centers | Pools | 13 |
| | 3.4 | Time po | ints and Visit Windows | 13 |
| 4 | Data A | Analysis | | 13 |
| | 4.1 | Populati | ons for Analysis | 14 |
| | | 4.1.1 | Subject Disposition | 14 |
| | | 4.1.2 | Protocol Deviations | 14 |
| | | 4.1.3 | Analysis Populations | 15 |
| | 4.2 | Subject | Demographics and Other Baseline Characteristics | 16 |
| | | 4.2.1 | Demographic Characteristics | 16 |
| | | 4.2.2 | General Medical History | 17 |
| | | 4.2.3 | Characteristics of Disease | 17 |
| | 4.3 | | ents (Study Product, Rescue Medication, other Concomitant es, Compliance) | 17 |
| | | 4.3.1 | Study Product Compliance and Exposure | |
| | | 4.3.2 | Prior and Concomitant Medication | |
| | 4.4 | Analysis | s of Efficacy | |
| | | 4.4.1 | Primary Efficacy Endpoint | |
| | | 4.4.2 | Secondary Efficacy Variables | |

| | | 4.4.3 | Handling of Missing Values/Censoring/Discontinuations | 25 |
|---|---|---|---|---|
| | 4.5 | Analysi | is of Secondary Objectives | 25 |
| | | 4.5.1 | Efficacy (Secondary) | 25 |
| | 4.6 | Explora | atory Analysis | 25 |
| | 4.7 | Analysi | is of Safety | 27 |
| | | 4.7.1 | Adverse Events and Serious Adverse Events | |
| | | 4.7.2 | Laboratory Tests | 27 |
| | | 4.7.3 | Vital Signs and Anthropometry | |
| | | 4.7.4 | Findings on Physical Examination | |
| | | 4.7.5 | Other Safety Variables | 28 |
| | 4.8 | Analysi | is of Other Variables | |
| 5 | Chan | • | Protocol Defined Statistical Analysis Plan | |
| 6 | | _ | Sables, Figures and Listings | |
| Att | - | | of Data Displays | |
| 7 | | | 1 7 | |

# **Abbreviations**

| AE | adverse event |
|--------|-----------------------------------------------|
| AGP | Alpha 1-acid glycoprotein |
| ANCOVA | Analysis of covariance |
| ANOVA | Analysis of variance |
| ARI | Acute respiratory illnesses |
| BMI | Body mass index |
| CRF | Case Report Form |
| CNS | Central Nervous System |
| CRP | C-reactive protein |
| CTCAE | Common Terminology Criteria for Adverse Event |
| DE | Design Effect |
| DF | Diagnosis Form |
| ENT | Ear, nose, throat |
| FSFV | First subject first visit |
| g | Gram |
| GI | Gastrointestinal |
| GSKCH | GlaxoSmithKline Consumer Healthcare |
| HAZ | Height for age Z score |
| НЬ | Hemoglobin |
| HBS | Human biological sample |
| IDDS | Individual Dietary Diversity Score |
| ITT | Intent to treat |
| LAR | Legally appropriate representative |
| LM | Lactulose; mannitol |

| MFC | Master formulation code |
|------|-----------------------------------------|
| mg | Milligram |
| mITT | Modified Intend to treat |
| ml | Milliliter |
| MMN | multiple micronutrient |
| MMRM | Mixed model repeated measure |
| MN | multiple nutrient |
| PP | per protocol |
| RAP | Reporting and Statistical Analysis Plan |
| RDA | Recommended Dietary Allowance |
| SAE | Serious adverse event |
| SD | Standard deviation |
| sIgA | Salivary immunoglobulin A |
| SOC | System Organ Class |
| SP | Study Physician |
| SPWR | Study Physician Weekly Review |
| sTfR | Serum transferrin receptor |
| WHO | World Health Organization |

The purpose of this Statistical Reporting and Analysis Plan is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 204477 version 5.0 dated 31October 2017.

# 1 Summary of Key Protocol Information

The purpose of this trial is to demonstrate the efficacy and safety of fortified malt based food on immunity outcomes in school children 7 to 10 years of age. Efficacy will be demonstrated as superiority of fortified malt based food on test vs. control group on the primary efficacy outcomes, number of ill days during nine months of intervention.

Safety will be demonstrated through assessment of adverse events (AEs).

# 1.1 Study Design

## **Overall Design**

This is a single centre, multiple sites, open label, two-arm, parallel-group, stratified by gender, matched pair cluster randomized, controlled study.

#### **Visit 1 - Screening Visit**

The following assessments will be conducted

- Informed consent and assent
- Demographics
- Medical history
- Current/concomitant medications
- General physical examination
- Vital signs
- Haemoglobin (Hb) assessment using Pronto
- Anthropometric measurements (height and weight)
- Inclusion/exclusion criteria evaluation
- Subject Eligibility

- 24 hr dietary recall & dietary diversity survey
- Parental/legally appropriate representative (LAR) training on the completion of the 'Symptom Check List'
- Dispense blank Parent/LAR Symptom Checklist and Product Compliance Report Forms

#### Visit 2 - Baseline Visit

The following assessments will be conducted

- Current/concomitant medications
- Continued eligibility criteria
- Sample collection for urinary Neopterin test & lactulose/mannitol test
- Sample collection for analysis of serum ferritin, serum transferrin receptor (sTfR), C-reactive protein(CRP), alpha 1-acid glycoprotein (AGP), salivary immunoglobulin A (sIgA) & nutritional biochemistry (for micronutrients vitamins A, B12, D, E, folate, and of the trace elements selenium, zinc, copper, and iron)
- AE monitoring

#### Visit 3, 4, 5, 6, 7, 8, 9, SPWR and Product Administration Visits

The following assessments will be conducted

- Current/concomitant medications
- Continued eligibility criteria
- Dietary counselling will be administered to all study participants and their parents/LARs.
- Test Group will be administered to all study participants in the test group.
- Study physician weekly review (SPWR) visits will be conducted on a weekly basis until End of Study Visit. Parent/LAR symptom checklist & Product Compliance Report Forms will be collected and reviewed.
- Adverse event(AE) monitoring

## Visit 10 - End of Study Visit

The following assessments will be conducted

- Current/concomitant medication
- General physical examination
- Vital signs
- Anthropometric measurements (height and weight)
- Continued eligibility criteria
- 24 hr dietary recall & dietary diversity survey
- Sample collection for urinary Neopterin test & lactulose/mannitol test
- Sample collection for analysis of serum ferritin, sTfR, CRP, AGP, sIgA & nutritional biochemistry (for micronutrients vitamins A, B12, D, E, folate, and of the trace elements selenium, zinc, copper, and iron)
- AE monitoring
- Study completion and medical sign-off

# 1.2 Study Objectives

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| To determine the total number of ill days due to GI and respiratory illnesses in participants receiving fortified malt based food (Test Group) with dietary counselling in comparison to participants receiving only dietary counselling over a period of nine months. | Total number of ill days due to<br>GI and respiratory illnesses. |
| Secondary Objectives | Secondary Endpoints |
| To compare the following variables in participants receiving the fortified malt based food (Test Group) along with dietary counselling to participants receiving only | • |

| | dietary counselling over a period of nine months. | | |
|---|---|---|---|
| • | Frequency of GI and respiratory illnesses. | • | Number of episodes of GI and respiratory illnesses. |
| • | Severity of GI and respiratory illnesses. | • | Severity of GI and respiratory illnesses. |
| • | School absenteeism due to GI and respiratory illnesses. | • | School absenteeism due to GI and respiratory illnesses. |
| • | Change from baseline (measured at screening) in body mass index (BMI). | • | BMI at screening and end of study. |
| • | Change from baseline in gut integrity/health as measured by Lactulose Mannitol test. | • | Gut integrity/health as measured by Lactulose Mannitol test at baseline and end of study. |
| • | Change from baseline in gut integrity/health as measured by Urinary Neopterin test. | • | Gut integrity/health as measured by Urinary Neopterin test at baseline and end of study. |
| • | Change from baseline in mucosal immunity as measured by Salivary Immunoglobulin A (IgA) status. | • | Salivary Immunoglobulin A (IgA) status at baseline and end of study. |
| • | Change from baseline in levels of micronutrients Vitamin A, B12, D (25-hydroxycholecalciferol), E, folate, of the trace elements selenium, zinc, copper, and iron as determined by blood draw and analysis. | • | Levels of micronutrients<br>Vitamin A, B12, D (25-<br>hydroxycholecalciferol), E,<br>folate, of the trace elements<br>selenium, zinc, copper, and<br>iron at baseline and end of<br>study. |
| • | Change from baseline levels of ferritin, | • | Levels of ferritin, sTfR, CRP, |

| serum transferrin receptor (sTfR), C-reactive protein (CRP), and Alpha 1-acid glycoprotein (AGP) as determined by blood draw and analysis. | and AGP at baseline and end of study. |
|---|---|
| Change from baseline (measured at screening) in dietary diversity score, assessed through 24-hour Individual Dietary Diversity Score (IDDS). | Dietary diversity score assessed through 24-hour IDDS at screening and end of study. |
| Change from baseline (measured at screening) in energy, protein, carbohydrates and fat consumption, assessed through 24-hour dietary recall survey. | Intake of energy, protein,<br>carbohydrate, and fat from 24-<br>hour dietary recall survey at<br>screening and end of study. |

#### 1.3 Treatments

The following product groups will be used for this study-

- Test group- Fortified malt based food plus dietary counselling
- Control group- Dietary counselling

# 1.4 Sample Size Calculation

The primary efficacy variable of the study is the total number of ill days due to GI and respiratory illnesses. The sample size has been calculated based on the assumption of an average of 7 ill days in the control group with a difference of 10% between the treatments.

Years Lost due to Disability (YLD) is a measure of the burden of disease from its morbidity. Below are data that are specific to India: As per the data from Global Burden Disease, WHO 2010 study (GBD, WHO, 2012; IHME, 2013) and Census India, 2011, YLD per child in the 5-9-year age group, due to diarrhea, LRTIs, other infectious disease and nutritional deficiencies is 8.274 days/child per year or 6.21 days/child per 9 months.

Thus, based on above data, approximately 7 ill days due to GI and respiratory illnesses per 9 months has been assumed in this proposed study population of 7-10 year olds.

The sample size is based on the primary endpoint. No sample size considerations have been taken into account for secondary objectives.

The simulated data were also used based upon the assumption of a Poisson distribution per study treatment. On observation of these simulated data, it was considered that these Poisson distributions were not heavily skewed and, as a result, normal distributions may be

assumed. Consequently, a normality assumption has been adopted for both the generation of sample size and the intended approach to the statistical analysis.

Because of assumption of Poisson distribution, estimates of variability were calculated as square root of mean.

Mean of control was assumed to be 7.0 and standard deviation (SD) was 2.65, mean of test group was 6.3 and SD was 2.51. To be able to achieve 80% power, 215 participants per treatment arm (Total = 430) will be required to complete the study in case of individual randomisation. This assumes 5% level of significance (two tailed t-test).

As this study is using cluster randomization, and design effect (DE) needs to be considered for sample size calculations. Scientific literature suggests, DE due to cluster sampling strategy can be assumed to be 1.5 [Rosner, B, 1986]. Same has been assumed in one study, which used three-stage systematic cluster sampling [Dandona R *et al*, 2008].

Using the following formula from Hemming et al, 2011:

$$N*=N \times DE$$

Where N\*=Number of participants required for cluster randomized trial

N = Number of participants required for individual randomization

DE = design effect

And assuming DE to be 1.5, the number of evaluable participants completing the study required would be 323 per arm (Total=646).

To allow for 30% drop-out rate, a total of 924 participants will be randomized.

Approximately 1300 participants will be screened to randomize approximately 924 participants in order to obtain 646 participants completing the study.

# 2 Planned Analyses

#### 2.1 Interim Analysis

No interim analysis is planned.

## 2.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants who have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and database has been locked.

3. All criteria for un-blinding the randomization codes have been met and the randomization codes have been distributed.

# 3 Considerations for data analyses and Data Handling Conventions

#### 3.1 Baseline Definition

For parameters height, weight, BMI, height for age Z score (HAZ), individual diversity dietary score (IDDS), carbohydrate, fat and energy from 24 hour dietary recall assessments conducted at screening visit will be considered as baseline and for all other endpoints the baseline value will be the latest pre-dose assessment Visit 2 with a non-missing value.

Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

# 3.2 Subgroups/Stratifications

To control for possible effects of gender, a balanced ratio of boys and girls in the test and the control groups will be targeted. The study will be stratified by gender to recruit a target ratio of 50% girls and 50% boys, with a minimum of 40% of either gender and a maximum of 60% of either gender.

#### 3.3 Centers Pools

This study is conducted in multiple (4) schools, with two schools in each product group.

# 3.4 Time points and Visit Windows

The time points and visits for this study are defined in the section "Schedule of Events" of the protocol. Any deviation from the study schedule will be reviewed case-by-case basis to determine whether the data should be excluded from the Per Protocol (PP) population. A time window non-compliance listing will be produced for the Blinded Data Review Meeting (BDRM) only.

# 4 Data Analysis

Data analysis will be performed by Syneos Health. The statistical analysis software used will be SAS Studio version 9.4 or higher.

Prior to database closure a BDRM will be conducted in which various aspects of the trial will be discussed and agreed.

Unless otherwise described below, all listings will be produced for enrolled population.

## 4.1 Populations for Analysis

Tables described in this section will be produced for enrolled population.

# 4.1.1 Subject Disposition

Screen failures are defined as participants who consented to participate in the study but were not subsequently enrolled (i.e., excluded basis inclusion/exclusion criteria). A summary of the number of participants screened and the number of screen failures with reasons of their exclusion will be presented (Table 14.1.1). Percentage of screen failure participants will be based on total number of screened participants. Subject disposition will also be summarized by product group and overall as the number and percentage of participants who completed the study, with the number who discontinue broken down by reason for discontinuation (Table 14.1.1). The table will also summarize the number and percent of participants assigned to each analysis population (refer to Section 4.1.3). The percentage will be based on total number of participants enrolled in each product group and overall.

Subject disposition including the participants status (completer, Yes/No), demographic data (age and race), screening date, product groups (including test product and dietary counselling) start date and time, the duration in the study or trial and the specific reason for discontinuation, will be listed for enrolled population (Listing 16.2.1.1) by product group.

Duration in the study or trial will be calculated using the formula below –

(Date of completion/withdrawal minus date of baseline visit)+1

Subject disposition information for non-enrolled participants will include subject number, demographic information (age and race), screening date, reason for screen failure and details if any regarding the reason for screen failure (Listing 16.2.1.2).

#### 4.1.2 Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study. Data will be reviewed prior to un-blinding and closure of the database to ensure all important deviations are captured and categorized. Participants with major protocol deviations (defined below) will be excluded from the PP population.

Major deviations of the protocol procedures identified as liable to influence the efficacy outcomes of the study may include, but will not be necessarily limited to the following:

- Violation of inclusion or exclusion criteria
- Significant non-compliance with assigned treatment
- Use of prohibited treatment or medication before or during the study
- Any other reason identified which may affect the efficacy assessments

The number and percentage of participants with any major protocol deviations will be presented by product group and overall (Table 14.1.2) and listed (Listing 16.2.2.1). Any minor protocol deviations will be listed similarly (Listing 16.2.2.2).

# 4.1.3 Analysis Populations

Six analysis populations are defined.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened<br>Subjects | All participants who enter the study and sign the informed consent form. This population includes screen failures as well. | Disposition, AE listing |
| Enrolled<br>Population | All participants who attended baseline visit will be considered in enrolled population. | Protocol deviations, AE, efficacy, demographic characteristic, disposition and medical history listings |
| Safety | Comprise of all participants who received at least one dose of study product (i.e. either only dietary counselling or both supplement and dietary counselling) during the study. | • Safety |
| | This population will be based on the product to which the participant was planned to receive. | |
| Intent-To-Treat (ITT) | All participants in the safety population with any post-treatment assessment (SPWR is considered as post-treatment assessment) will be included in Intent-to-treat (ITT) population. | • Efficacy |
| | This population will be based on the product to which the participant was planned to receive. | |
| Modified Intent-<br>To-Treat | • All participants in the ITT population who have completed entire study of 9 months | • Primary,<br>Secondary |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| (mITT) | (i.e., attended up to end study visit) will be included in modified intent-to-treat (mITT) population. | Exploratory<br>Efficacy |
| | This population will be based on the product to which the participant was planned to receive. | |
| Per-Protocol • Participants who have all post-treatment assessment and do not have any major protocol deviations that would affect efficacy assessments. | | • Efficacy |
| | Participants with major protocol deviations will be excluded. Depending on the nature of the major protocol deviation and impact on the efficacy variable (s), subjects will be either completely excluded from PP population or only partially excluded from the PP analyses. This will be determined on a case-by-case basis. | |

The primary population for assessment of efficacy will be the mITT Population. A PP analysis will be performed on the primary variable if more than 5 % of the subjects in the mITT Population are excluded from the PP Population.

Participants excluded from any of the analysis populations will be listed (Listing 16.2.3.1), with the reason for exclusion.

# 4.2 Subject Demographics and Other Baseline Characteristics

Demographic and baseline characteristics summaries will be produced for the Safety, ITT and mITT population.

## 4.2.1 Demographic Characteristics

Descriptive statistics (number of subjects [n], mean, and median, standard deviation [SD], minimum and maximum) for the continuous variables and frequency (n) and percentages (%) for categorical variables will be provided for demographic variables.

The continuous variable includes age (years), height (cm), weight (kg), BMI and HAZ and categorical variables include gender, race, and HAZ (for ranges:-3 to -2 and -2 to -1).

This data will be summarized descriptively for all participants in Safety (Table 14.1.4.1), ITT (Table 14.1.4.2), mITT (Table 14.1.4.3) and if required on the PP Population (Table 14.1.4.4). Demographic information will be listed (Listing 16.2.4.1) for enrolled population.

No formal statistical analysis will be performed for this data.

#### 4.2.2 General Medical History

Medical history data will be listed (Listing 16.2.4.2) with start date and end date or ongoing at the start of study product. A data listing will also be produced for evaluation of major protocol deviations at the blinded data review stage.

#### 4.2.3 Characteristics of Disease

Not Applicable.

# 4.3 Treatments (Study Product, Rescue Medication, other Concomitant Therapies, Compliance)

Compliance data will be summarized on the mITT population. Exposure and other medications will be listed on the enrolled population.

## 4.3.1 Study Product Compliance and Exposure

For doses administered at school, study-personnel will supervise and ensure complete consumption of test product.

The descriptive summary of total number of expected amount of product to be consumed, actual amount product consumed by product group and overall for all participants in mITT population (Table 14.2.1.1).

The compliance will be calculated using following formula –

#### **Test product compliance:**

Test product compliance = Actual Consumption X 100/Expected Consumption

Where, actual and expected consumption are defined below:

- Expected consumption = (2X 150 mL of drink X number of days\* between first and last treatment day in the study)
- Actual consumption = Expected consumption (xx mL total left over at morning + xx mL left over at evening)]

### **Dietary Counselling Compliance:**

<sup>\*</sup>up to maximum of 9 months (to be converted in days) (as test product is only administered maximum up to 9 month regardless last visit day in study)

The dietary counselling compliance will be calculated using following formulas:

#### • Participants:

- Compliance with Mandatory dietary counselling= (Number of sessions out of session numbers 1 or 2 attended by participant divided by 2) X 100
- O Compliance with Follow-up sessions dietary counselling= (Number of sessions out of session numbers 3-7 attended by participant divided by 5) X 100

#### • Parents/LAR:

- Compliance with Mandatory dietary counselling= (Number of sessions out of session numbers 1 or 2 attended by parents/LAR divided by 2) X 100
- o Compliance with Follow-up sessions dietary counselling= (Number of sessions out of session numbers 3-7 attended by parents/LAR divided by 5) X 100

Study product compliance listing (Listing 16.2.5.1) using enrolled population will be presented at the time of blinded data review process. Noncompliance will be assessed on a participant by participant basis. Those participants with product compliance less than 70% or non-compliant with dietary counselling will be excluded from the PP population. Any participant excluded from PP population will be clearly documented in the population definition document.

Exposure to the study product in days will be calculated as date of last day in the study minus date of first date of study product administration +1 for the test group.

Exposure to the study product in days will be calculated as date of last day in the study minus date of first date of dietary counselling +1 for the control group.

Exposure data will be listed (Listing 16.2.5.1) using enrolled population.

#### 4.3.2 Prior and Concomitant Medication

Prior or concomitant medication taken by or administered to a participant will be recorded in the case report form. The prior and concomitant medications will be coded using an internal validated medication dictionary, GSK Drug.

Prior medications are defined as those which stopped before the first administration of study product start date. If the stop date is unknown or incomplete and medication cannot be considered as stopped prior to first administration then the medication will be considered as concomitant medication.

Concomitant medications are defined as the medications ongoing on or after first study product start date.

Unknown dates will not be imputed, however if the start date is unknown, then it will be assumed to concomitant medication, unless the partial start date or stop date indicates differently.

Prior and concomitant medications/non-drug therapies will be listed by participant, with preferred term, indication, dose, dose form, frequency, route, start date, end date or ongoing and start day relative to first dose of study product (Listing 16.2.5.2 and Listing 16.2.5.3).

# 4.4 Analysis of Efficacy

## 4.4.1 Primary Efficacy Endpoint

## 4.4.1.1 Primary Efficacy Endpoint Definition

The primary efficacy variable of the study is the number of ill days over a period of nine months.

The definition of number of illness days is following –

**Number of illness days:** Number of days a subject is ill because of GI and/or respiratory illnesses as diagnosed by study physician, as per the criteria defined, over the intervention duration. This corresponds to total number of days (symptomatic or asymptomatic) in an episode of illness. Each episode is defined as each incidence of illness followed by at least 3 symptom free days.

In an episode if the first occurrence is due to GI illness and second occurrence is due to respiratory illness with less than 3 symptom free days then the overall episode due to GI and/or respiratory will be counted as one and separately it will be one each for GI and respiratory.

The asymptomatic days (or symptom free) days will be calculated programmatically based on the date mentioned on the Diagnosis Form in the following way –

Asymptomatic day = (Second occurrence start date - First occurrence end date) - 1

If asymptomatic day is less than 3 days then two occurrences of illnesses will be calculated and considered as single episode.

Else if asymptomatic days are greater than or equal to 3 days then two occurrences of illnesses will be calculated and considered as different episodes.

Descriptive statistics (n, mean, SD, SE, median, minimum and maximum) by product group will be provided (Table 14.2.2.1). Number of ill days due to GI and/or respiratory illnesses will be listed for each subject (Listing 16.2.6.18).

## 4.4.1.2 Statistical Hypothesis, Model, and Method of Analysis

For the primary variable, primary analysis will be performed on participants on the mITT population.

The null hypothesis of interest is:

H0: There is no difference between the numbers of illness days for the product groups.

The alternative hypothesis of interest is:

H1: There is a difference in between the numbers of illness days for the product groups.

The number of ill days will be analysed using the analysis of variance (ANCOVA) model. The ANCOVA will have cluster (school) as a random effect, product group and gender as fixed effects and baseline IDDS as a covariate.

Adjusted means, 95% confidence intervals (CI), within product group p-values for each product group, product group difference, intracluster correlation, 95% confidence interval of the difference and the between-product group p-values based on the statistical model described above will also be presented (Table 14.2.2.2).

All statistical tests of hypotheses will be two-sided and will employ a level of significance of  $\alpha = 0.05$ .

The simulated data used for the sample size calculations were based upon the assumption of a Poisson distribution per product group. However, on observation of these simulated data, it was considered that these Poisson distributions were not heavily skewed and, as a result, normal distributions may be assumed. Consequently, a normality assumption has been adopted for both the generation of sample size and the intended approach to the statistical analysis.

However, the assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation (for example, log or square root or Poisson regression using Proc Genmod) or by performing appropriate non-parametric tests (e.g., Van Elteren, rank ANCOVA).

#### 4.4.1.3 Supportive Analyses

As a part of sensitivity analysis a Mixed Model Repeated Measure (MMRM) model will be used. MMRM model will be just an analysis including multiple visits with defined structure of correlation among visits. In this study unstructured covariance matrix will be used. The number of ill days will be analysed using model with cluster (school) as a random effect; product group, gender, and visit and (product group and visit) interaction as fixed effects and baseline IDDS as a covariate.

This will be conducted on the primary efficacy endpoints on the ITT population (Table 14.2.2.2a).

#### 4.4.2 Secondary Efficacy Variables

The analysis of secondary efficacy variables will be on the mITT population.

The secondary efficacy variables are:

#### • Frequency of GI and Respiratory illness

Frequency of GI and respiratory illnesses defined as total number of illness episodes of GI and/or respiratory illnesses, divided by duration of intervention in month, where each episode is defined as each incidence of illness followed by at least 3 symptom free days will be summarized in a table for the product groups (Table 14.2.3.1).

The frequency of GI and respiratory illnesses will be calculated as following –

Frequency (per month) = No of episodes X 30/ Number of days between first (BV) and last visit

Frequency of GI and respiratory illnesses will be analysed together using analysis of covariance (ANCOVA) model. The model will include cluster (school) as a random effect; fixed effects for product group and gender; and baseline IDDS as a covariate. Adjusted means, 95% confidence intervals, intracluster correlation, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model described above will also be presented (Table 14.2.3.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation or by performing sensitivity analysis or by appropriate non-parametric tests (e.g., Van Elteren, rank ANCOVA).

#### • Analysis on Severity of GI and Respiratory illness:

Frequency and percentages of severity episodes of GI and respiratory illnesses will be summarized in a table together and also separately (Table 14.2.4.1). If an episode comprises of occurrences of different severities, then the highest severity will be considered as the overall severity. Severity grades will be displayed in the tables for the GI and respiratory illness as mentioned in the Appendix 5 of the Protocol version 5.0.

Frequencies of severity (Mild, moderate, or severe) episode between product groups will be compared using Chi-Square test (if frequencies are greater than 5%). If frequencies are  $\leq 5\%$  in any product group, then these will be compared using Fisher's exact test between product groups (Table 14.2.4.1).

### • Analysis of School absenteeism due to GI and Respiratory illness:

Descriptive statistics (n, mean, and median, SD, minimum and maximum) will be provided for school absenteeism due to GI and respiratory illnesses (Table 14.2.5.1).

School absenteeism due to GI and respiratory illnesses will analysed together using analysis of variance (ANCOVA) model. The model will include cluster (school) as a random effect; fixed effects for product group and gender; and baseline IDDS as a covariate.

Adjusted means, 95% confidence intervals, within product group p-values for each product group, product group difference, intracluster correlation, 95% confidence interval of the difference and the between-product group p-values based on the statistical model described above will also be presented (Table 14.2.5.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation or by performing appropriate non-parametric tests (e.g., Van Elteren, rank ANCOVA).

#### • Analysis of Body Mass Index (BMI):

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) will be provided for BMI (Table 14.2.6.1). Change from baseline of BMI will be analysed using an analysis of covariance (ANCOVA) model. The model will include cluster (school) as a random effect; fixed effects for product group and gender; baseline BMI assessment recorded at screening visit and baseline IDDS as a covariate. Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model described above will also be presented (Table 14.2.6.2). The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation or by performing appropriate non-parametric tests (e.g., Van Elteren).

# • Analysis of Gut integrity/health as measured by Lactulose: Mannitol test and Urinary Neopterin test:

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) for the Lactulose: Mannitol and Urinary Neopterin will be provided in a table (Table 14.2.7.1). Change from baseline in gut integrity/health as measured by Lactulose: Mannitol test and Urinary Neopterin test and will be analysed using an ANCOVA model.

The model will include cluster (school) as a random effect; fixed effects for product group and gender, baseline guts integrity/health assessment as a covariate. Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model described above will also be presented (Table 14.2.7.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation or by performing appropriate non-parametric tests (e.g., Van Elteren).

#### • Analysis of Salivary IgA (sIgA):

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) for the sIgA will be provided (Table 14.2.8.1). Change from baseline of sIgA will be analysed using an ANCOVA model. The model will include cluster (school) as a random effect; fixed effects for product group and gender; baseline sIgA assessment as a covariate. Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model will also be presented (Table 14.2.8.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation (eg., log or square root) or by performing appropriate non-parametric tests (e.g., Van Elteren).

In case of logarithm transformation log base 10 will be used and additionally geometric mean will be provided for the descriptive statistics.

#### • Analysis of Micronutrients from blood sample:

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) for the micronutrients (Vitamin A, B12, D (25 Hydroxy calciferol), E, folate, of the trace elements selenium, zinc, copper, and iron) concentration levels will be provided (Table 14.2.9.1).

Change from baseline in concentration levels of micronutrients (Vitamin A, B12, D (25 Hydroxy calciferol), E, folate, of the trace elements selenium, zinc, copper, and iron) will be analysed using an ANCOVA model. The model will include cluster (school) as a random effect; fixed effects for product group and gender; baseline assessments concentration levels and baseline IDDS as a covariate.

Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model will also be presented (Table 14.2.9.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation (eg., log or square root) or performing appropriate non-parametric tests (e.g., Van Elteren).

In case of logarithm transformation log base 10 will be used and additionally geometric mean will be provided for the descriptive statistics.

#### • Analysis of serum variables from blood sample:

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) for the serum parameters (ferritin, serum-transferrin receptor (sTfR), C-reactive protein (CRP), and Alpha 1-acid glycoprotein (AGP)) will be provided (Table 14.2.10.1). Change from baseline in concentration levels of serum parameters C-reactive protein (CRP), and Alpha 1-acid glycoprotein (AGP)) will be analysed using an ANCOVA model.

The model will include cluster (school) as a random effect; fixed effects for product group and gender; baseline assessments of each serum concentration levels as a covariate. Also, a separate ANCOVA model will be used to analyse change from baseline ferritin, serum-transferrin receptor (sTfR), with cluster (school) as a random effect; product group and gender as fixed effects and baseline assessment concentration levels, CRP and AGP concentration levels as covariates.

Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model will also be presented (Table 14.2.10.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation (eg., log or square root) or by performing appropriate non-parametric tests (e.g., Van Elteren).

In case of logarithm transformation log base 10 will be used and additionally geometric mean will be provided for the descriptive statistics.

#### • Analysis of Individual Dietary Diversity Score (IDDS):

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) for the IDDS will be provided (Table 14.2.11.1). Also, change from baseline IDDS will be presented in a summary table by product group. Change from baseline in dietary diversity score will be analysed using an ANCOVA model. The model will include cluster (school) as a random effect; fixed effects for product group, and gender; baseline assessments at screening as a covariate.

Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model will also be presented (Table 14.2.11.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation (eg., log or square root) or by performing appropriate non-parametric tests (e.g., Van Elteren).

IDDS categories are defined as below –

- 1.  $\leq$  3 food groups Lowest dietary diversity
- 2. 4 and 5 food groups Medium dietary diversity
- 3.  $\geq$  6 food groups High dietary diversity

Frequency and percentages for each category of IDDS will also be presented (Table 14.2.11.3).

Frequencies for each category between product groups will be compared using Chi-Square test (if frequencies are greater than 5%). If frequencies are  $\leq$  5% in any product group, then these will be compared using Fisher's exact test between product groups (Table 14.2.11.3).

# Analysis of energy, protein, carbohydrate and fat from 24-hour dietary recall survey:

Descriptive statistics (n, mean, and median, SD, SE, minimum and maximum) for the Energy, Protein, Fat and Carbohydrate will be provided (Table 14.2.12.1).

Change from baseline of each assessment will be analysed using the ANCOVA model with cluster (school) as a random effect; product group and gender as fixed effects; baseline assessments for each responses as a covariate.

Adjusted means, intracluster correlation, 95% confidence intervals, within product group p-values for each product group, product group difference, 95% confidence interval of the difference and the between-product group p-values based on the statistical model will also be presented (Table 14.2.12.2).

The assumptions of normality and homogeneity of variance will be investigated and violation of these assumptions may be overcome using suitable transformation (eg., log or square root) or by performing appropriate non-parametric tests (e.g., Van Elteren).

## 4.4.3 Handling of Missing Values/Censoring/Discontinuations

Missing endpoints data will not be imputed, only subjects that completed the study are included on the mITT population.

#### 4.5 Analysis of Secondary Objectives

# 4.5.1 Efficacy (Secondary)

Refer Section 4.4.2 for the analysis of secondary objectives.

# 4.6 Exploratory Analysis

#### • Analysis of number of ill days over 3 and 6 months:

The number of ill days due to GI and respiratory illnesses over 3 months and 6 months separately on the ITT population who have completed the study for 3 months and 6 GlaxoSmithKline Consumer Healthcare Confidential

months will be summarized and analyzed using the same model as used in the primary analysis (Table 14.2.13.1.1 and Table 14.2.13.1.2).

 Analysis of total number of ill days for GI and respiratory illness separately over 3, 6 and 9 months:

Primary analysis and the above analysis will be repeated for total number of ill days for GI and respiratory illness separately at months 3, 6 and 9 based on the ITT population (Table 14.2.13.2.1 and Table 14.2.13.2.2 for GI illness) and (Table 14.2.13.3.1 and Table 14.2.13.3.2 for respiratory illness).

• Analysis of total number of ill days due to GI and respiratory illnesses, school absenteeism (days), frequency (per month), severity by gender at 9 months:

It will be summarized and analysed and presented as detailed for the primary and secondary endpoint respectively by gender (Table 14.2.13.4.1 and Table 14.2.13.4.2 for ill days due to GI and respiratory illnesses), (Table 14.2.13.7.1 and Table 14.2.13.7.2 for school absenteeism (days)), (Table 14.2.13.5.1 and Table 14.2.13.5.2 for frequency (month)) and severity of episodes (Table 14.2.13.6.1).

• Analysis of change from baseline of HAZ, Height and Weight:

Change from baseline in HAZ, height and weight will be summarised and analysed using the same ANCOVA model as mentioned for the BMI analysis (Table 14.2.13.8.1 and Table 14.2.13.8.2 for HAZ), (Table 14.2.13.9.1 and Table 14.2.13.9.2 for height), (Table 14.2.13.10.1 and Table 14.2.13.10.2 for weight).

• Association between Gut integrity/health as measured by Lactulose: Mannitol test and Urinary Neopterin test with blood chemistry:

Correlation between micronutrients (Vitamin A, B12, D (25 Hydroxy calciferol), E, folate, selenium, zinc, copper, and iron) and gut integrity/health as measured by Lactulose: Mannitol test and Urinary Neopterin test will be computed at baseline and at visit 10 (Table 14.2.13.11,), Also, correlation between change from baseline micronutrients (Vitamin A, B12, D (25 Hydroxy calciferol), E, folate, selenium, zinc, copper, and iron) and change from baseline in gut integrity/health as measured by Lactulose: Mannitol test and Urinary Neopterin will be computed at month 9 (Table 14.2.13.12).

• Summary of Number of Ill Days Due to GI Illness and respiratory illnesses and separately by School over Month 3, 6 and 9:

Descriptive statistics tables for number of Ill days due to GI and Respiratory Illnesses by School (Table 14.2.14.1), number of Ill days due to GI Illnesses by School (Table 14.2.14.2) and number of Ill days due to Respiratory Illnesses by School (Table 14.2.14.3) will be presented.

# 4.7 Analysis of Safety

#### 4.7.1 Adverse Events and Serious Adverse Events

All safety data will be reported for the Safety Population as per planned study product received. The safety profile of the study product will be assessed with respect to AEs. All AEs will be reviewed by the Clinical Research Scientist or Designee prior to database freeze and will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

AEs will be regarded as treatment-emergent (TE) if they occur on or after the first study product administration. If this date is missing a suitable alternative will be used e.g. date of visit 3. All other AEs prior to this will be considered non-treatment emergent.

AEs will be regarded as treatment emergent for the control group if they occur on or after the first dietary session or visit 3.

The following summary tables and listings will be presented by product group.

- Table of Treatment Emergent Adverse Event (TEAEs) by System Organ Class and Preferred Term (Table 14.3.1.1)
- Table of TEAEs related to study treatment by System Organ Class and Preferred Term (Table 14.3.1.2)
- Table of TEAEs by System Organ Class, Preferred Term and Severity (Table 14.3.1.3)
- Listing of all AEs (Listing 16.2.7.1 for enrolled population; Listing 16.2.7.2 for non-enrolled subjects)
- Listing of death occurring during treatment (if any) will be listed by product group, including the date and study day of death, and the principal cause of death (Listing 14.3.2.1)
- Listing of non-fatal serious adverse events (Listing 14.3.2.2)
- Listing of TEAEs leading to withdrawal (Listing 14.3.2.3)

#### 4.7.2 Laboratory Tests

Laboratory parameters for which reference ranges will be available will be categorized with respect to reference ranges as: High, Low, Normal and Missing. The shift will be calculated with respect to reference ranges from baseline for the subsequent visits.

Laboratory results at baseline, and at month 9 will be presented in shift tables (Tables 14.3.5.3 - 14.3.5.17).

Laboratory normal ranges will be listed in Listing (Listings 16.2.6.17) and all laboratory test results will be listed in Listings (Listings 16.2.6.1 - 16.2.6.16).

#### 4.7.3 Vital Signs and Anthropometry

Vital signs heart rate (beats/min), and oral temperature (°F), height (cm), weight (kg), body mass index (kg/m²) and anthropometric parameter HAZ will be collected at screening and at month 9.

Observed values at each visit and change from baseline at post-baseline visit will be summarized on the safety population descriptively (n, mean, SD, SE, median, minimum, and maximum) by product group (Table 14.3.5.1).

All vital signs will be listed (Listing 16.2.9.1).

## 4.7.4 Findings on Physical Examination

The findings on the physical examination (Central Nervous System (CNS), Eyes, Ear Nose Throat (ENT), Respiratory, Cardiovascular, Gastrointestinal, Musculoskeletal, Neurological, Endocrine and Metabolic, Dermatological, Haematopoietic/Lymphatic) performed at screening, and month 9, will be listed (Listing 16.2.9.2).

## 4.7.5 Other Safety Variables

Hemoglobin (g/dL) collected at screening visit will be summarized descriptively for all subjects in safety population.

Observed values at screening visit will be summarized descriptively (n, mean, SD, SE, median, minimum, and maximum) by product group (Table 14.3.5.2).

Hemoglobin measurements will be listed (Listing 16.2.9.3).

#### 4.8 Analysis of Other Variables

Not applicable.

# 5 Changes to the Protocol Defined Statistical Analysis Plan

Any changes from the originally planned statistical analysis specified in the protocol (Dated: 10 October 2017) are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan |
|----------|---------------------------|
|----------|---------------------------|

| Statistical<br>Analysis<br>section | Statistical Analysis Plan | Rationale for Changes |
|---|---|---|
| • 4.1.3 | <ul><li>Enrolled population defined</li><li>Modified ITT population defined</li></ul> | Since this study uses cluster randomization<br>and not individual participant's randomized<br>so randomized population cannot be<br>defined. Instead enrolled population defined. |
| | | To allow the exclusion of some enrolled participants in a justified way (such as participant who were deemed ineligible after enrolment or certain participants who never started treatment). |
| • 4.4.1<br>and<br>4.4.2 | Primary, secondary and exploratory analysis will be done on mITT population. | Primary analysis should be done on participants those who are presented entire study duration. |
| | | Secondary and exploratory outcome data<br>(particularly those involving analysis on<br>human biological samples), are available<br>only after End of study visit (visit 10). |
| | | ANOVA model for analysis of ferritin, serum-<br>transferrin receptor (sTfR), is modified. |
| • 9.2.1 | PP analysis will be performed in case<br>there is a 5% difference observed<br>between number of subjects in mITT<br>(instead of ITT) and PP. | This change has been incorporated since<br>mITT is primary population of analysis |
| • 9.3.5 | The following analysis was removed | It will be part of potential post-hoc analysis |
| | Total number of ill days (GI and respiratory illnesses), number of episodes (GI and respiratory illnesses), and severity of GI and respiratory illnesses by screening, end of study, and change from baseline in DDS, energy, protein, carbohydrate and fat. | decided after study un-blinding if imbalances between product groups are observed for the variables. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical<br>Analysis<br>section | Statistical Analysis Plan | Rationale for Changes |
| <ul><li>9.3.2</li><li>9.3.3</li><li>9.3.5</li></ul> | Baseline IDDS has been added in the statistical model as covariate for the primary, secondary and other analysis since baseline IDDS has an impact on these analyses. | Morbidities are the important endpoints (both primary and secondary) in this study and scientific evidences suggest that these outcomes are associated with dietary diversity score (Oduor et al., 2013) (Kiboi et al., 2016). Also, factors such as nutritional and socioeconomic status which play important role in immunity status of children are also associated with dietary diversity. Dietary diversity is associated with socioeconomic status and household food security (Hoddinot & Yohannes, 2002; Hatloy et al., 2000). IDDS has been validated for several age/sex groups as proxy measures for macro and/ or micronutrient adequacy of the diet (FAO guidelines dietary diversity, 2011). Thus, the background diet is a major possible confounder in this nutritional intervention study. It thus becomes pertinent that confounding due to dietary intake measured through IDDS is controlled during statistical analysis. |

## • RAP Amendment 1

This RAP Amendment 1 provides details of modified analyses requested from the analysis described in the Statistical Reporting and Analysis Plan (final version 1.0). The section below provides a summary of the analysis with the justification for the request.

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical<br>Analysis<br>section | Statistical Analysis Plan | Rationale for Changes |
| <ul><li>9.3.2</li><li>9.3.3</li></ul> | For all ANCOVA analyses, "cluster (school)" will be included as a random | Handling "cluster" as random effect would avoid over-parametrisation and would allow for intracluster correlation. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical<br>Analysis<br>section | Statistical Analysis Plan | Rationale for Changes |
| • 9.3.5 | effect instead of a fixed effect. Present the estimate of the intra cluster correlation in the ANCOVA tables. | Adjusting for the intracluster correlation is necessary for a valid analysis. |

# 6 Template for Tables, Figures and Listings

This is a guideline which will give the guidance of product group labels that will be used for the table header and in the figures, listings and in the footnotes.

The product group labels for the column headings will be as follow:

Test Group and Control Group;

The product group comparison will be:

• Test Group vs Control Group

The order of the product groups will be following-

• 1st: Test Group

• 2nd: Control Group

In all the outputs following footnote will be added –

Test Group: Fortified malt based food + Dietary Counselling

Control Group: Dietary Counselling

# **Attachment 1: List of Data Displays**



#### Fortified malt based food

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

Table 14.1.1

**Subject Disposition** 

All Screened Subjects

Study Population: All Screened Subjects (N=xxx)

| | Test Group | Control Group | Overall |
|-----------------------------|------------|---------------|------------|
| | n (%) | n (%) | n (%) |
| TOTAL SUBJECTS SCREENED | | | xxx |
| SUBJECTS NOT ENROLLED | | | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | | | xxx (xx.x) |
| ADVERSE EVENT | | | xxx (xx.x) |
| SUBJECTS ENROLLED | xxx | xxx | xxx |
| COMPLETED STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT COMPLETE STUDY | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DID NOT MEET STUDY CRITERIA | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ADVERSE EVENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| LOST TO FOLLOW-UP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PROTOCOL VIOLATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| WITHDRAWAL OF CONSENT | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| OTHER | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

#### Fortified malt based food

#### 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| | Test Group | Control Group | Overall |
|-------------------|------------|---------------|------------|
| | n (%) | n (%) | n (%) |
| SAFETY POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ITT POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| mITT POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PP POPULATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Percentages for not enrolled category are based on number of screened subjects; percentages for enrolled category are based on number of enrolled subjects.

Program: xxxxxx.sas Source: Filename Page x of y

#### Fortified malt based food

204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Table 14.1.2

Incidence of Major Protocol Deviations

**Enrolled Population** 

Study Population: Enrolled (N=xxx)

| | Test Group | Control Group | Overall |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| SUBJECTS WITH AT LEAST ONE MAJOR PROTOCOL DEVIATION | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MAJOR PROTOCOL DEVIATIONS NOT LEADING TO EXCLUSION FROM PP | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| MAJOR PROTOCOL DEVIATIONS LEADING TO EXCLUSION FROM PP All VISITS | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| VISIT Y | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| DEVIATION REASON 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Test Group: Fortified malt based food + Dietary Counselling; Control Group: D | pietary Counselling | | |
| Program: xxxxxx.sas | Source: Filename | | Page x of y |

**Programming Note:** This table will list all major protocol deviations as defined in the population definition document.
# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

#### Table 14.1.4.1

#### **Demographic and Baseline Characteristics**

#### Safety Population

Study Population: Safety Population (N=XXX)

| | Test Group | Control Group | Overall |
|-----------------------------------|------------|---------------|------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| RACE n (%) | | | |
| AFRICAN AMERICAN/AFRICAN HERITAGE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| AMERICAN INDIAN OR ALASKAN NATIVE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| AGE (YEARS) | | | |
| n | xx | XX | xx |
| MEAN | xx.x | XX.X | XX.X |
| HAZ category n (%) | | | |
| ≥-3 to <-2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ≥-2 to ≤-1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| SEX n (%) | | | |
| FEMALE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GlaxoSmithKline Consumer Healthcare Confidential


# Fortified malt based food 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| | Test Group | Control Group | Overall |
|-------------------------|------------|---------------|------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| MALE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| HEIGHT (cm) | | | |
| n | xx | xx | хх |
| MEAN | xxx.xx | xxx.xx | XXX.XX |
| Height for age Z score | | | |
| n | xx | xx | XX |
| MEAN | xxx.xx | xxx.xx | XXX.XX |
| WEIGHT (kg) | | | |
| n | xx | xx | XX |
| MEAN | xxx.xx | xxx.xx | XXX.XX |
| BODY MASS INDEX (kg/m²) | | | |
| n | xx | xx | xx |
| MEAN | xxx.xx | xxx.xx | xxx.xx |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Percentages are based on number of subjects in each product group and overall.

| Fortified malt based food |
|---|
| 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018 |
| <b>Programming Note:</b> For continuous variables the summary statistics: n, Mean, SD, SE, Median, Minimum and Maximum will be displayed Similar table will be displayed for ITT population and mITT population. |

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.1.1

#### Study Product Compliance

#### Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

| | Statistics | Test Group | Control Group |
|---|---|---|---|
| | | (N = xxx) | (N = xxx) |
| TEST PRODUCT COMPLIANCE | | | |
| | n | xx | |
| | MEAN | x.xxx | |
| | SD | x.xxxx | |
| | MEDIAN | x.xxx | |
| | MINIMUM | x.xx | |
| | MAXIMUM | x.xx | |
| DIETARY COUNSELLING COMPLIANCE – MANDATORY SESSIONS | | | |
| PARTICIPANTS | n | xx | xx |
| | MEAN | x.xxx | x.xxx |
| | SD | x.xxxx | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | x.xx | x.xx |
| | MAXIMUM | x.xx | x.xx |
| PARENTS/LAR | n | xx | xx |

GlaxoSmithKline Consumer Healthcare Confidential


# Fortified malt based food 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| | Statistics | Test Group | Control Group |
|---|---|---|---|
| | | (N = xxx) | (N = xxx) |
| | MEAN | x.xxx | x.xxx |
| | SD | x.xxxx | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | x.xx | x.xx |
| | MAXIMUM | x.xx | x.xx |
| ETARY COUNSELLING COMPLIANCE FOLLOW-UP SESSIONS | | | |
| PATICIPANTS | n | xx | xx |
| | MEAN | x.xxx | x.xxx |
| | SD | x.xxxx | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | x.xx | x.xx |
| | MAXIMUM | x.xx | x.xx |
| PARENTS/LAR | n | xx | xx |
| | MEAN | x.xxx | x.xxx |
| | SD | x.xxxx | x.xxxx |
| | MEDIAN | x.xxx | x.xxx |
| | MINIMUM | x.xx | x.xx |
| | MAXIMUM | x.xx | x.xx |

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Statistics | Test Group | Control Group |
|------------|------------|---------------|
| | (N = xxx) | (N = xxx) |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Percentage is based on number of subjects in each product group.

Test product compliance = (actual consumption/expected consumption)\*100

Dietary Counselling Compliance:

Participants

Compliance with Mandatory dietary counselling= (Number of sessions out of session numbers 1 or 2 attended by participant divided by 2) X 100

Compliance with Follow-up sessions dietary counselling= (Number of sessions out of session numbers 3-7 attended by participant divided by 5) X 100

Parents/LAR:

Compliance with Mandatory dietary counselling= (Number of sessions out of session numbers 1 or 2 attended by Parents/LAR divided by 2) X 100

Compliance with Follow-up sessions dietary counselling= (Number of sessions out of session numbers 3-7 attended by Parents/LAR divided by 5) X 100

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.2.1

#### Summary of Number of Ill Days Due to GI and Respiratory Illnesses over Month 3, 6 and 9

#### Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

| Visit | Statistics | Test Group | Control Group | Overall |
|---------|------------|----------------|----------------|----------------|
| | | (N = xxx) | (N = xxx) | (N = xxx) |
| | | Observed Value | Observed Value | Observed Value |
| MONTH 3 | n | xxx | xxx | xxx |
| | MEAN | xx.xx | XX.XX | xx.xx |
| | SD | xx.xxx | xx.xxx | xx.xxx |
| | SE | x.xx | x.xx | x.xx |
| | MEDIAN | x.xx | x.xx | x.xx |
| | MINIMUM | xx.x | xx.x | xx.x |
| | MAXIMUM | XX.X | XX.X | xx.x |
| MONTH 6 | n | xxx | xxx | |
| | MEAN | xx.xx | xx.xx | |
| | SD | xx.xxx | xx.xxx | |
| | SE | x.xx | x.xx | |
| | MEDIAN | x.xx | x.xx | |

GlaxoSmithKline Consumer Healthcare Confidential


# Fortified malt based food 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Visit | Statistics | Test Group | Control Group | Overall |
|---------|------------|------------|---------------|-----------|
| | | (N = xxx) | (N = xxx) | (N = xxx) |
| | MINIMUM | xx.x | XX.X | |
| | MAXIMUM | xx.x | xx.x | |
| MONTH 9 | n | xxx | xxx | |
| | MEAN | xx.xx | xx.xx | |
| | SD | xx.xxx | xx.xxx | |
| | SE | x.xx | x.xx | |
| | MEDIAN | x.xx | x.xx | |
| | MINIMUM | xx.x | xx.x | |
| | MAXIMUM | xx.x | XX.X | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** Similar table will be generated for secondary and exploratory variables. For the exploratory analysis the similar table will be repeated including month 3, and month 6 using ITT population who completed month 3 and month 6.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.2.2

#### Statistical Analysis of Number of III Days Due to GI and Respiratory Illnesses at Month 9

#### Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

| | | | | | | | | Compa | arison with Control Grou | р |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Group | N | Adjusted Mean | SE | 95% CI | P-Value | Intracluster | Difference (SE) | 95% CI | P-Value |
| | | | | | | | Correlation | | | |
| MONTH 9 | Test Group | xxx | xx.xx | XX.XXX | xx.xx, xx.xx | 0.xxxx | x.xxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| | Control Group | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Analysis was performed using ANCOVA model with cluster (school) as a random effect; product group and gender as fixed effects and baseline IDDS as covariate.

Difference is Test Group minus Control Group such that a negative difference favors the Test Group.

Intracluster correlation performed on complete model.

Confidence interval (CI) are presented as calculated (not truncated) and could present also negative values. Such negative values within CI no to be used for result interpretations.

Program: xxxxxxx.sas Source: Filename Page x of y

# **Programming Note:**

- 1. This table is for the primary end point.
- 2. For the exploratory analysis the similar table will be repeated including month 3, and month 6 using ITT population who completed month 3 and month 6.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.2.2a

Statistical Analysis of Number of III Days Due to GI and Respiratory Illnesses using Repeated Measure at Month 9

#### Intent-to-Treat Population

Study Population: Intent-to-Treat Population (N = xxx)

| | | | | | | | | Compariso | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Group | N | Adjusted Mean | SE | 95% CI | P-Value | Intracluster | Difference (SE) | 95% CI | P-Value |
| | | | | | | | Correlation | | | |
| MONTH 9 | Test Group | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | x.xxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| | Control Group | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Analysis was performed using MMRM model with cluster (school) as a random effect; product group, gender, visit and (product group and visit) interaction as fixed effects and baseline IDDS as covariate.

Difference is Test Group minus Control Group such that a negative difference favors the Test Group.

Intracluster correlation performed on complete model.

Confidence interval (CI) is presented as calculated (not truncated) and could present also negative values. Such negative values within CI no to be used for result interpretations.

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** Similar table will be generated for all primary endpoints using imputed missing data. Direction of the difference should be with respect to the parameter which will be analyzed and should be checked with Clinical Research and Statistician for finalization.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol: 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.4.1

#### Summary and Statistical Analysis on Severity Episodes of GI and Respiratory Illnesses

#### Modified Intent-to-Treat Population

Study Population: Modified Intent to Treat Population (N=XXX)

| PREFERRED TERM | Test Group (N=XXX) | Control Group | P-VALUE[1] | P-VALUE[2] |
|---|---|---|---|---|
| SEVERITY | | (N=XXX) | | |
| GI ILLNESS | | | | |
| MILD | xx (xx.x) | xx (xx.x) | 0.xxx | 0.xxx |
| MODERATE | xx (xx.x) | xx (xx.x) | | |
| SEVERE | xx (xx.x) | xx (xx.x) | | |
| DIARRHOEA | | | | |
| MILD | xx (xx.x) | xx (xx.x) | 0.xxx | 0.xxx |
| MODERATE | xx (xx.x) | xx (xx.x) | | |
| SEVERE | xx (xx.x) | xx (xx.x) | | |
| VOMITTING | | | | |
| MILD | xx (xx.x) | xx (xx.x) | 0.xxx | 0.xxx |
| MODERATE | xx (xx.x) | xx (xx.x) | | |
| SEVERE | xx (xx.x) | xx (xx.x) | | |

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| PREFERRED TERM SEVERITY | Test Group (N=XXX) | Control Group<br>(N=XXX) | P-VALUE[1] | P-VALUE[2] |
|---|---|---|---|---|
| RESPIRATORY ILLNESS MILD | xx (xx.x) | xx (xx.x) | 0.xxx | 0.xxx |
| MODERATE | xx (xx.x) | xx (xx.x) | | |
| SEVERE | xx (xx.x) | xx (xx.x) | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

[1] p-value is from the Chi-Square test.

[2] p-value is from the Fisher's exact test.

The numbers are based on the episodes with worst severity.

Program: xxxxxx.sas Source: Filename Page x of y

**Programming note:** The table will represent on the episodes

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

Table 14.2.6.1

Summary of BMI (kg/m2)

#### Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

| Visit | Statistics | Т | est Group | Cont | trol Group | O | verall |
|---|---|---|---|---|---|---|---|
| | | (N = xxx) | | 1) | V = xxx | (N | = xxx) |
| | | Observed Value | Change from Baseline | Observed Value | Change from Baseline | Observed Value | Change from Baseline |
| SCREENING | n | xxx | | xxx | | | xxx |
| | MEAN | xx.xx | | xx.xx | | : | xx.xx |
| | SD | xx.xxx | | xx.xxx | | х | x.xxx |
| | SE | x.xx | | x.xx | | | x.xx |
| | MEDIAN | x.xx | | x.xx | | | x.xx |
| | MINIMUM | xx.x | | xx.x | | | xx.x |
| | MAXIMUM | xx.x | | xx.x | | | xx.x |
| MONTH 9 | n | xxx | xxx | xxx | | | |
| | MEAN | xx.xx | xx.xx | xx.xx | | | |
| | SD | XX.XXX | xx.xxx | xx.xxx | | | |
| | SE | x.xx | x.xx | x.xx | | | |

GlaxoSmithKline Consumer Healthcare Confidential


204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Visit | Statistics | Test Group<br>(N = xxx) | | Control Group | Overall |
|---|---|---|---|---|---|
| | | | | (N = xxx) | (N = xxx) |
| | _ | | | | |
| | MEDIAN | x.xx | X.XX | x.xx | |
| | MINIMUM | XX.X | xx.x | xx.x | |
| | MAXIMUM | xx.x | xx.x | XX.X | |
| Test Group: Fortified m | alt based food + Dietary Counselli | ng; Control Group: [ | Dietary Counselling | | |
| Program: xxxxxx.sas | | | Source: Filename | 2 | Page x of y |

**Programming Note:** Similar table will be generated for all secondary variables. For the parameters Lactulose: Mannitol test and Urinary Neopterin test, Salivary IgA, micronutrients, ferritin, serum-transferrin receptor (sTfR), C-reactive protein (CRP), and Alpha 1-acid glycoprotein (AGP), energy, protein, carbohydrate and fat the first visit will be the visit 2 baseline visit.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.6.2

#### Statistical Analysis of BMI (kg/m²) Change from Baseline at Month 9

#### Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

| | | | | | | | | Comparison with Control Group | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Group | N | Adjusted Mean | SE | 95% CI | P-Value | Intracluster | Difference (SE) | 95% CI | P-Value |
| | | | | | | | Correlation | | | |
| MONTH 9 | Test Group | XXX | XX.XX | xx.xxx | xx.xx, xx.xx | 0.xxxx | x.xxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| | Control Group | XXX | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Analysis was performed on change from baseline BMI using ANCOVA model with cluster (school) as a random effect; product group and gender as fixed effects; and baseline BMI and IDDS as covariate.

Difference is test group minus control group such that a positive difference favors the test group.

Intracluster correlation performed on complete model.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol: 204477 Program Run Date: DDMMMYYYY

#### Table 14.2.11.3

#### Summary and Statistical Analysis on Individual Dietary Diversity Score (IDDS) Categories

#### Modified Intent-To-Treat Population

Study Population: Modified Intent to Treat Population (N=XXX)

| IDDS Category | Test Group | Control Group | P-VALUE[1] | P-VALUE[2] |
|-------------------|------------|---------------|------------|------------|
| | (N=XXX) | (N=XXX) | | |
| LOWEST DIVERSITY | xx (xx.x) | xx (xx.x) | | |
| MEDIUM DIVERSITY | xx (xx.x) | xx (xx.x) | 0.xxx | 0.xxx |
| HIGHEST DIVERSITY | xx (xx.x) | xx (xx.x) | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

IDDS: Individual Dietary Diversity Score

[1] p-value is from the Chi-Square test.

[2] p-value is from the Fisher's exact test.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### 14.2.13.4.1

Summary of Number of Ill Days Due to GI and Respiratory Illnesses by Gender at Month 9

Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

<By Variable >: XXXXXX (N = xxx)

| Visit | Statistics | Test Group | Control Group | Overall |
|---------|------------|----------------|----------------|----------------|
| | | (N = xxx) | (N = xxx) | (N = xxx) |
| | | Observed Value | Observed Value | Observed Value |
| MONTH 9 | n | xxx | xxx | |
| | MEAN | XX.XX | xx.xx | |
| | SD | XX.XXX | xx.xxx | |
| | SE | x.xx | x.xx | |
| | MEDIAN | x.xx | x.xx | |
| | MINIMUM | xx.x | xx.x | |
| | MAXIMUM | xx.x | xx.x | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### 14.2.13.4.2

#### Statistical Analysis of Number of III Days Due to GI and Respiratory Illnesses by Gender at Month 9

#### Modified Intent-to-Treat Population

Study Population: Modified Intent-to-Treat Population (N = xxx)

<By Variable >: XXXXXX (N = xxx)

| | | | | | | | | Comparison with Control Group | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Group | N | Adjusted Mean | SE | 95% CI | P-Value | Intracluster | Difference (SE) | 95% CI | P-Value |
| | | | | | | | Correlation | | | |
| MONTH 9 | Test Group | XXX | XX.XX | xx.xxx | xx.xx, xx.xx | 0.xxxx | x.xxx | xx.xx (xx.xxx) | xx.xx, xx.xx | 0.xxxx |
| | Control Group | xxx | xx.xx | xx.xxx | xx.xx, xx.xx | 0.xxxx | | | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Analysis was performed using ANCOVA model with cluster (school) as a random effect; product group and gender as fixed effects and baseline IDDS as covariate.

Difference is Test Group minus Control Group such that a negative difference favors the Test Group.

Intracluster correlation performed on complete model.

Confidence interval (CI) is presented as calculated (not truncated) and could present also negative values. Such negative values within CI no to be used for result interpretations.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol: 204477 Program Run Date: DDMMMYYYY

Table 14.2.13.11

Correlation between Blood Chemistry and Gut Integrity Health by Lactulose: Mannitol and Urinary Neopterin Test by Time Point

Modified Intent-To-Treat Population

Study Population: Modified Intent-to-Treat Population (N=XXX)

Time point: Baseline

| | Test | Group | | Contro | l Group |
|---|---|---|---|---|---|
| | (N | =xx) | | (N=xx) | |
| | Lactulose Mannitol | Urinary<br>Neopterin Test | | Lactulose<br>Mannitol | Urinary<br>Neopterin Test |
| Vitamin A | XX.X | xx.x | Vitamin A | XX.X | xx.x |
| Vitamin B12 | xx.x | xx.x | Vitamin B12 | xx.x | xx.x |
| Vitamin D | xx.x | xx.x | Vitamin D | xx.x | XX.X |
| Vitamin E | xx.x | xx.x | Vitamin E | xx.x | xx.x |
| Folate | XX.X | xx.x | Folate | xx.x | xx.x |
| Selenium | xx.x | xx.x | Selenium | xx.x | xx.x |
| Zinc | XX.X | xx.x | Zinc | XX.X | xx.x |
| Copper | XX.X | xx.x | Copper | xx.x | xx.x |
| Iron | xx.x | xx.x | Iron | xx.x | xx.x |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** The same structure will be in the next page for MONTH 9

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol: 204477 Program Run Date: DDMMMYYYY

Table 14.3.1.1

### Treatment Emergent Adverse Event by System Organ Class and Preferred Term

Safety Population

Study Population: Safety Population (N=xxx)

| System Organ Class | Test Gr | oup | Control | Group | Overa | II |
|---|---|---|---|---|---|---|
| Preferred Term | (N = xxx) | | (N = xxx) | | (N = xxx) | |
| | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE AE | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| NUMBER OF SUBJECTS WITH NO AE | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC 1 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| PT 1 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| PT 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| SOC 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| PT 1 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| PT 2 | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |

GlaxoSmithKline Consumer Healthcare Confidential

204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| System Organ Class | Test Gr | Test Group | | l Group | Overall | |
|---|---|---|---|---|---|---|
| Preferred Term | (N = x | (N = xxx) | | = xxx) | (N = xxx) | |
| | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| Test Group: Fortified malt based food + Dietary C | Counselling; Control Group: Dietary Counse | ling | | | | _ |
| n (%) = Number (percent) of subjects; nAE = Num | ber of adverse events. | | | | | |

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** Similar table will be generated for treatment related adverse events.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Table 14.3.1.3

#### Treatment Emergent Adverse Event by System Organ Class, Preferred Term and Severity

Safety Population

Study Population: Safety Population (N=xxx)

| System Organ Class | Severity | Test | Group | Cont | Control Group | | Overall |
|---|---|---|---|---|---|---|---|
| Preferred Term | | (N : | (N = xxx) | | (N = xxx) | | (N = xxx) |
| | | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| System Organ Class 1 | Mild | xx (xx.x) | XX | xx (xx.x) | xx | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| Preferred Term 1 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| Preferred Term 2 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |
| | Severe | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | xx |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

n (%) = Number (percent) of subjects; nAE = Number of adverse events.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Statistics

Protocol 204477 Program Run Date: DDMMMYYYY

Test Group

#### Table 14.3.5.1

#### Summary of Vital Signs and Anthropometry Parameters

#### Safety Population

Control Group

Overall

Study Population: Safety Population (N = xxx)

Parameter: <Parameter Name (Unit)>

Visit

| | | (N = | xxx) | 1) | N = xxx) | (N = xxx) |
|---|---|---|---|---|---|---|
| | | Observed Value | Change from Baseline | Observed Value | Change from Baseline | Observed Value |
| SCREENING | n | XXX | | xxx | | xxx |
| | MEAN | xxx.x | | xxx.x | | xxx.x |
| | SD | xxx.xx | | xxx.xx | | xxx.xx |
| | SE | xxx.xx | | xxx.xx | | xxx.xx |
| | MEDIAN | xxx.x | | xxx.x | | xxx.x |
| | MINIMUM | xxx | | xxx | | xxx |
| | MAXIMUM | Xxx | | Xxx | | Xxx |
| MONTH 9 | n | xxx | xxx | xxx | XXX | |
| | MEAN | xxx.x | xxx.x | xxx.x | xxx.x | |
| | SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | |
| | SE | xxx.xx | xxx.xx | xxx.xx | XXX.XX | |

GlaxoSmithKline Consumer Healthcare Confidential


204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Visit | Statistics | Test Group | | Contro | ol Group | Overall |
|-------|------------|------------|-----------|---------|----------|-----------|
| | | (N = | (N = xxx) | | = xxx) | (N = xxx) |
| | MEDIAN | xxx.x | xxx.x | xxx.x | xxx.x | |
| | MINIMUM | xxx | xxx | xxx | xxx | |
| | MAXIMUM | Xxx Xxx | | Xxx Xxx | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** This table will continue for all other scheduled visits and for all vital signs [Height (cm), Weight (kg), BMI (kg/m2), Heat rate (beats/min), Height for age Z score, and Oral body temperature (°F)]. Display overall only for the baseline visit.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMMYYYY

#### Table 14.3.5.3

Shift Table for Lactulose: Mannitol Test and Urinary Neopterin Test (unit)

#### Safety Population

Study Population: Safety Population (N = xxx)

Parameter: <Parameter (Unit)>, Reference range: <xx-xx>

| | | | | Test Group | | | | | Control Group | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Baseline | | | | | Baseline | | |
| Visit | Result | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) | Total<br>n (%) | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| | Low | and the control | | 201 (011) | NO (10 / 10 | NO. (NO. 14) | NA 604 N | NO. (10.) 10 | and the control | and have a | 20/00/20 |
| Baseline | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | | | | | | | | | | |
| | High | | | | | | | | | | |
| | Missing | | | | | | | | | | |
| | Total | | | | | | | | | | |
| Month 9 | Low | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Normal | | | | | | | | | | |
| | High | | | | | | | | | | |
| | Missing | | | | | | | | | | |
| | Total | | | | | | | | | | |

204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| | | Test Group | | | | | Control Group | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | | | Baseline | | | | | Baseline | | |
| | Result | Low | Normal | High | Missing | Total | Low | Normal | High | Missing | Total |
| Visit | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | , | V/ | (, | (/ | (, | , | , | , | , | |

Low, normal, and high categories defined by reference ranges.

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** This table will continue for all other scheduled visits and laboratory parameters

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

#### Listing 16.1.7

#### Randomization Information

| School Number | School Name | Randomization Number | Product Group |
|---------------|-------------|----------------------|---------------|
| xxxxxx | | XXXXXX | |

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.1.1

Subject Disposition

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| School<br>Number | Subject<br>Number | Age/ Sex<br>/Race [1] | Screening Date | Study Product Start<br>Date and Time | Last Study Product<br>Administration Date<br>and Time | Date of<br>Completion or<br>Withdrawal | Duration in the<br>Study (days) [2] | Completed<br>the Study | Primary Reason for<br>Withdrawal | Further Details [3] |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XX/A1 | DDMMMYYYY | DDMMMYYYY:HH:MM | DDMMMYYYY:HH:MM | DDMMMYYYY | XXX | Yes | | |
| XXXXXX | XXXXXX | XX/A6 | DDMMMYYYY | DDMMMYYYY:HH:MM | DDMMMYYYY:HH:MM | DDMMMYYYY | XXX | No | Other | XXXXXX |
| xxxxx | XXXXXX | XX/A4 | DDMMMYYYY | DDMMMYYYY:HH:MM | DDMMMYYYY:HH:MM | DDMMMYYYY | | | | |

Test Product: Fortified malt based food + Dietary Counselling; Control Product: Dietary Counselling

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple.

<sup>[2]</sup> Duration in the study = (Date of completion/withdrawal minus date of baseline visit)+ 1

<sup>[3]</sup> Further details of reasons for withdrawal.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.1.2

Subject Disposition

Non-Enrolled Population

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple.

<sup>[2]</sup> Further details of reasons for screen failure.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.2.1

**Major Protocol Deviations** 

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject Number | Age/Sex/Race [1] | Visit(s)Excluded from PP Population | Deviation Reason |
|---|---|---|---|
| 10001 | 25/I | All | Did not meet Inclusion criteria |
| | | From Visit 3 | Inclusion criteria |
| | | Visit 4 only | Treatment non-compliance |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** This listing is based on details in the population definition document.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Protocol 204477 | Program Run Date: DDMMYYYY |
|-----------------|----------------------------|
|-----------------|----------------------------|

Listing 16.2.2.2

Minor Protocol Deviations

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject Number | Age/Sex/Race [1] | Deviation Sequence | Start Date/Time of<br>Deviation | End Date/Time of Deviation | Deviation Description |
|---|---|---|---|---|---|
| XXXXXX | XX/A1 | 1 | DDMMMYYYY:HH:MM | DDMMMYYYY:HH:MM | XXXXXX |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Protocol 204477 | Program Run Date: DDMMYYYY |
|-----------------|----------------------------|
|-----------------|----------------------------|

Listing 16.2.3.1

**Exclusion from Analysis Populations** 

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject Number | Age/Sex/Race[1] | Safety Population | ITT Population | mITT Population | PP population |
|---|---|---|---|---|---|
| XXXXXX | XX/A1 | YES | YES | YES | YES |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

[1] Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = Multiple

Program: xxxxxx.sas Source: Filename Page x of y

Programming Note: This listing is based on population definition document.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

#### Listing 16.2.4.1

#### **Demographic and Baseline Characteristics**

#### **Enrolled Population**

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject<br>Number | Age (years) | Sex | Race | Height (cm) | Weight (kg) | Body Mass Index<br>(kg/m²) | Height for age Z score |
|---|---|---|---|---|---|---|---|
| XXXXXX | XX | Female | African American/African Heritage | xxx.x | xxx.x | xx.x | |
| XXXXXX | XX | Female | African American/African Heritage | xxx.x | xxx.x | xx.x | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.4.2

Medical History

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject Number | Age/Sex/Race[1] | Any Medical History | Medical Condition | Start Date | End Date or Ongoing |
|---|---|---|---|---|---|
| xxxxxx | XX/A1 | Yes | xxxxxx | DDMMMYYYY | DDMMMYYYY |
| XXXXXX | XX/A6 | Yes | XXXXXX | DDMMMYYYY | Ongoing |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT = multiple

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Protocol 20 | 7192 | | | | | | | | | Program Run Date: DDM | 1MYYYY |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Li | sting 16.2.5.1 | | | | |
| | | | | | | Study Product Ac | lministration and Co | mpliance | | | |
| | | | | | | Enro | olled Population | | | | |
| Study Popu | lation: Enr | olled Populat | tion (N=xx) | | | | | | | | |
| Product Gro | oup: Test G | Group | | | | | | | | | |
| Subject<br>Number | Age/<br>Race | Visit | Exposure[<br>2] | Expected amount of drink | Actual<br>Amount of | Test Group<br>Compliance | Dietary Counsel | ling Complianc | e | | |
| | [1] | | | to be<br>consumed[3] | Drink<br>Consumed | (%)[5] | | | | | |
| | | | | | [4] | | Mandatory sess compliance [6] | ion | | sion compliance<br>and parents)[7] | |
| | | | | | | | Participants | Parents/L<br>AR | -<br>Participants | Parents/LAR | |
| XXXXXX | XX/A<br>1 | Overall | | | | | | | | | |
| | | Overall | | х | x | 98 | | | | | |

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

- [1] Age in years; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White White/Caucasian/European Heritage, MT = multiple.
- [2] Exposure for test group: date of last day in the study date of first date of test group administration +1; Exposure for control group: date of last day in the study date of first date of dietary counselling +1.
- [3] Expected consumption = 2X 150 mL of drink X number of days between first and last treatment day in the study
- [4] Actual consumption = [Expected consumption (xx mL total left over at morning + xx mL left over at evening)]
- [5] Test product compliance in %= (actual consumption/ expected consumption) X 100
- [6] Mandatory sessions compliance by both participants and patents=( Number of sessions out of session numbers 1 or 2 attended by participant/ parents divided by 2) X 100
- [7] Compliance with Follow-up sessions dietary counselling= (Number of sessions out of session numbers 3-7 attended by participant and/or parents/LAR divided by 5) X 100

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.5.2

**Prior Medications** 

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject<br>Number | Age/Sex/Race[1] | Sequence<br>Number | Drug Name<br>[GSK Drug Synonym] | Reason for<br>Medication | Route of Admin. | Dose per Admin.<br>(unit) | Frequency | Start Date (Study Day [2]) | End Date/ Ongoing |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XX/A6 | 1 | xxxxxx<br>[xxxxxx] | XXXXXX | xxxxxx | XXXXXX (xx) | xxxxxx | DDMMMYYYY<br>(XX) | Ongoing |
| xxxxxx | XX/A6 | 1 | XXXXXX<br>[XXXXXX] | XXXXXX | xxxxxx | XXXXXX (xx) | xxxxxx | DDMMMYYYY<br>(XX) | DDMMMYYYY |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

**Programming Note:** Similar listing will be generated for Concomitant Medications and Non-Drug Therapies.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

<sup>[2]</sup> Study day relative to the date of first date of dietary counselling.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.6.1

Urine Neopterin Assay

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject<br>Number | Age/Sex<br>/Race<br>[1] | Visit | Date of<br>Visit | Was<br>Assessment<br>Performed? | Date of Sample<br>Collection/Time<br>of Sample<br>Collection | Normal<br>Range | Panic<br>Range | Result<br>(unit) | Abnormality<br>[2] | Change<br>from<br>Baseline | Comment |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XX/N | Scree<br>ning | DDMMMY<br>YYY | Yes | | xx.x-xx.x | xx.x-<br>xx.x | xx.x | L | | xxx |
| | | Baseli<br>ne | DDMMMY<br>YYY | | | | | xx.x | Н | | ххх |
| | | Visit 5 | DDMMMY<br>YYY | Yes | | | | xx.x | CS | xx.x | XXXX |
| | | Visit 6 | DDMMMY<br>YYY | | | | | | | xx.x | |

## **Programming Note:**

• Repeat the same layout for listing 16.2.6.2-16.2.6.16

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

#### Listing 16.2.6.17

#### Listing of Normal Range for Saliva Blood and Urine Parameters

| Parameter (Unit) | Biological Matrix | Gender | Age Range (in years) | Normal Ra | ange | Panic | Range |
|---|---|---|---|---|---|---|---|
| | | | _ | Lower Limit | Upper Limit | Lower Limit | Upper Limit |
| Serum Type I Collagen Cross-<br>inked C-telopeptide (unit) | Blood | Male | хх-хх | | | | |
| | | Female | XX-XX | | | | |

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Protocol 204477 | Program Run Date: DDMMYYYY |
|-----------------|----------------------------|
|-----------------|----------------------------|

Listing 16.2.6.18

Listing of Diagnosis Data

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Product

| Subject Number | Age/Sex/R<br>ace[1] | Sequence Number | Diagnosis | Start Date | End Date | Severity | School Absenteeism (No. of days in this week) |
|---|---|---|---|---|---|---|---|
| xxxxxx | XX/N | | Vomiting | 31MAR2018 | DDMMMYYYY | Mild | No |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage.

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.7.1

All Adverse Events

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject<br>Number | Age/Sex/R<br>ace[1] | Adverse Event (Preferred Term) | Start Date/Time/<br>Study Day[2] | End Date/<br>Time | Frequency/<br>Intensity | Related to<br>Study<br>Product? | Action Taken<br>with Study<br>Product | Outcome | Serious? | Subject<br>Withdrawn |
|---|---|---|---|---|---|---|---|---|---|---|
| | | [System Organ Class] | | | | | | | | |
| XXXXXX | XX/N | HEADACHE | 31MAR2017/ | DDMMMYYYY/ | SINGLE | No | NOT | RECOVERED/ | NO | NO |
| | | (NERVOUS SYSTEM<br>DISORDER) | HH:MM:SS/ 3 | HH:MM:SS | EPISODE/<br>MILD | | APPLICABLE | RESOLVED | | |
| | | [xxxxxx] | | | | | | | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxxx.sas Source: Filename Page x of y

## Programming Note for Listing 16.2.7.2:

- Repeat the same layout for listing 16.2.7.2
- Population should be used 'Non randomized Subjects'
- The fourth column should be only 'Start Date/Time (take out Study Day)'
- Delete the footnote related to study day and adjust the numbers accordingly.

GlaxoSmithKline Consumer Healthcare Confidential

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage.

<sup>[2]</sup> Study day relative to the date of first date of dietary counselling

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.9.1

Vital Signs and Anthropometry Parameter

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject | Age/Sex | Visit | Date of | Date of | Height (cm) | | Weight (Kg) | | Heart | | Oral Tempe | rature (F) | Height for ag | ge Z score |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | /Race[1] | | Visit | Assessment | | | | | Rate (beats/min) | | | | | |
| | | | | | Observed value | Change<br>from<br>Baseline | Observed value | Change<br>from<br>Baseline | Observed value | Change<br>from<br>Baseline | Observed value | Change from<br>Baseline | Observed<br>value | Change from<br>Baseline |
| | | Screening | DDMMM<br>YYYY | DDMMMYYYY | | | | | | | | | | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

[1] Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

Program: xxxxxx.sas Source: Filename Page x of y

Programmer Note: Please also include information for Body Mass Index (kg/m²) prior to Height (cm)

## 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

Protocol 204477 Program Run Date: DDMMYYYY

Listing 16.2.9.2

**Physical Examination** 

**Enrolled Population** 

Study Population: Enrolled Population (N=xx)

Product Group: Test Group

| Subject Number | Age/Sex Race[1] | Visit | Date of Visit | Body System | Finding | Description of Abnormality, CS or Not Examined |
|---|---|---|---|---|---|---|
| XXXXXX | XX/N | Screening | DDMMMYYYY | CNS | Normal | |
| | | | | Eyes | Normal | |
| | | | | ENT | Abnormal, CS | xxxxxx |
| | | | | Respiratory | Normal | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

Program: xxxxxx.sas Source: Filename Page x of y

Programming Note for Listing 16.2.9.2: If subjects has abnormality description and CS description, please concatenate both separating with ','.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

# 204477 Statistical Reporting and Analysis Plan Amendment 1 2 November 2018

| Protocol 20 | )4477 | | | | | | Program Run Date: DDMMYYYY |
|---|---|---|---|---|---|---|---|
| | | | | | Listing 16.2.9.3 | | |
| | | | | | Hemoglobin Assessment | | |
| | | | | | <b>Enrolled Population</b> | | |
| | Study Popul | ation: Enrolled Populatio | n (N=xx) | | | | |
| | Product Gro | | | | | | |
| | Subject<br>Number | Age/Sex/Race | Visit | Date of Visit | Was Hb Assessment Performed? | Hb Assessment Results (g/dL) | |
| | Number | [1] | | | | | |
| | | | | | | Observed value | |
| | XXXXXX | XX/N | Screening | DDMMMYYYY | Yes | | |
| | | | Baseline | DDMMMYYYY | | XX.X | |
| | | | | | | XX.X | |
| | | | Visit 5 | DDMMMYYYY | Yes | | |
| | | | Visit 6 | DDMMMYYYY | | XX.X | |

Test Group: Fortified malt based food + Dietary Counselling; Control Group: Dietary Counselling

[1] Age in years; Sex: F = Female, M = Male; Race: A1 = African American/African Heritage, A2 = American Indian Or Alaskan Native, A3 = Asian-Central/South Asian Heritage, A4 = Asian-East Asian Heritage, A5 = Asian-Japanese Heritage, A6 = Asian-South East Asian Heritage, N = Native Hawaiian Or Other Pacific Islander, W1 = White-Arabic/North African Heritage, W2 = White - White/Caucasian/European Heritage, MT=Multiple.

Program: xxxxxx.sas Source: Filename Page x of y

GlaxoSmithKline Consumer Healthcare Confidential


## 7 References

- 1. Oduor, Francis Odhiambo. Malnutrition, dietary diversity, morbidity and associated factors among schoolchildren in Kibwezi district, Kenya. Diss. University of Nairobi, 2013.
- 2. Kiboi, Willy Kahanya. Dietary diversity, nutrient intake and nutritional status among pregnant women in Laikipia county, Kenya. Diss. Kenyatta University, 2016
- 3. Ruel MT (2003). Is dietary diversity an indicator of food security or dietary quality? A review of measurement issues and research needs. Food Nutr Bull 24: 231–232.
- 4. Hoddinott, J and Yohannes, Y. (2002). Dietary diversity as a food security indicator. FANTA 2002, Washington DC. http://www.aed.org/Health/upload/dietarydiversity.pdf
- 5. Hatloy, A., Hallund, J., Diarra, MM and Oshaug A. (2000). Food variety, socioeconomic status and nutritional status in urban and rural areas in Koutiala (Mali). Public Health Nutrition 3:57-65.
- 6. Food and Agriculture Organization (FAO) Guidelines for measuring household and individual dietary diversity. Rome, Italy: Food and Agriculture Organization of the United Nations; 2011.
- 7. Dandona R, Kumar GA, Ameer MA, Ahmed GM, Dandona L. Incidence and burden of road traffic injuries in urban India. Inj Prev. 2008 Dec;14(6):354-9. Available from <a href="http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2777413/pdf/ukmss-28072.pdf">http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2777413/pdf/ukmss-28072.pdf</a>
- 8. Hemming Karla, Alan J Girling, Alice J Sitch, Jennifer Marsh and Richard J Lilford. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Medical Research Methodology 2011, 11:102, 1471-2288.
- 9. Rosner, B. Fundamentals of Biostatistics. 2nd edition. PWS Publishers; Boston: 1986. p. 84-92.p. 302-68.p. 404-8.
- 10. Global Burden of Disease (GBD) at WHO, 2012.